CLINICAL TRIAL: NCT04254861
Title: Regenerative Treatment of Intrabony Defects With GTR and PRGF: A Randomised, Single-blind, Parallel-group Clinical Trial
Brief Title: Autologous Platelet Concentrate (APC) in Intrabony Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS Project ID: 259229; COCR0021 (Other: CORC)
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Periodontal Diseases
Keywords: Intrabony defect; Periodontitis; PRGF
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Intervention Model Description: This is a randomized, single-blind, parallel-group controlled trial comparing the efficacy of GTR and PRGF ENDORET® in the treatment of periodontal intrabony defects. The trial will follow the recommendations of the Consolidated Standards of Reporting Trials (CONSORT) statement.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, both participants and clinicians performing the surgical intervention will be unblinded. Conversely, outcome examiners will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simplified Papilla Preservation Flap (SPPF) and PRGF (Experimental)
  Interventions: Procedure: Simplified Papilla Preservation Flap (SPPF) and PRGF ENDORET (PRGF ENDORET®-KMU16)
- Simplified Papilla Preservation Flap (SPPF) and GTR (Active Comparator)
  Interventions: Procedure: Simplified Papilla Preservation Flap (SPPF) and GTR

INTERVENTIONS:
Procedure: Simplified Papilla Preservation Flap (SPPF) and PRGF ENDORET (PRGF ENDORET®-KMU16) — A simplified papilla preservation flap (SPPF) will be performed. The clot phase of PRGF ENDORET (F2) will be placed in the defect, while the fibrin membrane phase (F1) will cover it.
  Blood will be extracted and collected in dedicated tubes and then centrifuged. Up to 8 tubes of 9ml will be extracted. The time from the start of the extraction to the start of the centrifugation of the tubes must not exceed 4mins.
  After centrifugation, the blood is separated into three components: Plasma rich in growth factors, White cells or leukocytes, red blood cells: this is the red column occupying the bottom of the tube.
  Following BTI's instructions, fractioning of the centrifuged blood will be performed in order to separate Fraction 2 (F2), which contains a greater number of platelets and growth factors and will be used as a clot inside the periodontal defect from Fraction 1 (F1), which will be used as a fibrin member to cover the clot. The flaps will be repositioned and sutured.
  Other Names: Simplified Papilla Preservation Flap (SPPF) and GTR
  Arms: Simplified Papilla Preservation Flap (SPPF) and PRGF
Procedure: Simplified Papilla Preservation Flap (SPPF) and GTR — A simplified papilla preservation flap (SPPF) will be performed. The defect will then be treated according to the guided tissue regeneration (GTR) principle (control group). A deproteinized bovine bone mineral (DBBM) graft will be placed in the defect and covered by a collagen membrane.
  Arms: Simplified Papilla Preservation Flap (SPPF) and GTR

SUMMARY:
The aim of this 12-month clinical study is to treat patients affected by gum disease (periodontitis) by a minor gum surgery that aims to reduce the depth of the gum pockets. In particular, the study will compare two types of gum surgery, one based on the use of a product derived from the patients' own blood (PRGF, platelet autologous concentrate), and the other based on the use of an animal-derived bone graft and membrane that have been in the market for the past 30 years. Both procedures aim to regenerate bone and gum tissue that is damaged by the disease. 74, ≥ 25-year-old, otherwise healthy, patients affected by gum disease will be recruited at the Barts and The London Dental Hospital. Participants will be randomly (by chance) assigned to receive one of the two treatments. Throughout the study, we will assess gum's health by taking some measurements around teeth and gums. In addition, we will use non-invasive technologies to assess changes in temperature, blood flow and face's swelling at different time-points. Patients will be given specific questionnaires to evaluate their preferences and the impact that each surgical treatment had in their everyday life. One intra-oral x-ray will be performed before the surgery and after 12 months to assess if new bone has formed around the teeth involved in the surgery, as per standard procedure.

DETAILED DESCRIPTION:
This is a randomized, single-blind, parallel-group controlled trial comparing the efficacy of GTR and PRGF ENDORET in the treatment of periodontal intrabony defects. The trial will follow the recommendations of the Consolidated Standards of Reporting Trials (CONSORT) statement.

No negative control (SPPF alone) has been considered for this project since several studies have demonstrated that guided tissue regeneration (GTR) associated or not with bone grafts results in better clinical outcomes than access flap alone in the treatment of periodontal intrabony defects.

The study consists of 9 visits over a minimum period of 13 months and will take place at the Centre for Oral Clinical Research (COCR), at the Institute of Dentistry, Barts and The London School of Medicine and Dentistry, Queen Mary University of London.

Visit 1 - Baseline -

* Informed consent, medical/dental history and demographics
* Record concomitant medications and smoking history
* Height and weight measurement
* Standardised peri-apical x-ray in the area selected for the study
* Periodontal assessment by a blind and calibrated examiner, consisting of full mouth PPD, REC, BOP, mobility and furcation involvement will be recorded. PPD, REC, plaque and BOP will be recorded at 6 sites per tooth.
* Intra-oral 3D scan in the area selected for the study
* PROMs assessment (OIDP, and Global ratings of Periodontal Health and Quality of Life, EuroQoI-5D-5L)
* 3D extra-oral morphometric and Thermal scan
* Laser speckle contrast imaging, LSCI
* Pre-treatment hygiene phase, including supragingival scale and polish of all teeth and oral hygiene instructions
* Randomization to one of the two treatment groups by the study co-ordinator. The treatment allocation will be concealed in an opaque envelope. A treatment visit will be scheduled within the following 6 weeks.

Visit 2 - Surgical intervention - (within 6 weeks from Visit 1)

* Query to update medical/dental history and record adverse events and/or concomitant medications
* Recording of the number of defect walls
* Study treatment according to randomization (PRGF ENDORET or GTR)
* Intra-oral 3D scan in the area selected for the study (scan taken immediately after surgery)
* Record of surgery time
* Post-surgical instructions
* 3D extra-oral morphometric and thermal scan (scan taken immediately after surgery)

Visit 3 - 2 days follow-up - (2 days ±1 days from Visit 2)

* Query to update medical/dental history and record adverse events and/or concomitant medications
* Visual assessment of gingival healing and recording of early healing index (EHI)
* Laser speckle contrast imaging, LSCI
* Intra-oral 3D scan in the area selected for the study
* 3D extra-oral morphometric and Thermal scan
* PROMs assessment (Evaluation of global changes in quality of life and evaluation of patient perception about therapy)

Visit 4 - Suture removal - (7 days +3 days from visit 2)

* Query to update medical/dental history and record adverse events and/or concomitant medications
* Visual assessment of gingival healing and recording of early healing index (EHI)
* Laser speckle contrast imaging, LSCI
* Intra-oral 3D scan in the area selected for the study
* 3D extra-oral morphometric and Thermal scan
* Suture removal
* Supra-gingival polishing and reinforcement of oral hygiene instructions
* PROMs assessment (Evaluation of global changes in quality of life and evaluation of patient perception about therapy)

Visit 5 - 2 weeks follow up visit- (14 days ±3 days from visit 2)

* Query to update medical/dental history and record adverse events and/or concomitant medications
* Visual assessment of gingival healing and recording of early healing index (EHI)
* Laser speckle contrast imaging, LSCI
* Intra-oral 3D scan in the area selected for the study
* 3D extra-oral morphometric and thermal scan
* Supra-gingival polishing and reinforcement of oral hygiene instructions
* PROMs assessment (Evaluation of global changes in quality of life and evaluation of patient perception about therapy)

Visit 6 - 4 weeks follow up visit- (28 days ±3 days from visit 2)

* Query to update medical/dental history and record adverse events and/or concomitant medications
* Visual assessment of gingival healing
* Intra-oral 3D scan in the area selected for the study
* 3D extra-oral morphometric and Thermal scan
* Supra-gingival polishing and reinforcement of oral hygiene instructions
* PROMs assessment (Global ratings of Periodontal Health and Quality of Life, Evaluation of global changes in quality of life, and Eevaluation of patient perception about therapy and EuroQoI-5D-5L)

Visit 7 - 3 months follow up visit- (3 months ±7 days from visit 2)

* Query to update medical/dental history and record adverse events and/or concomitant medications
* Recording of PPD, REC, BOP, PI and mobility on the tooth involved in the surgical intervention and 2 adjacent teeth by a blind and calibrated examiner
* PROMs assessment (OIDP, Global ratings of Periodontal Health and Quality of Life, and eEvaluation of global changes in quality of life and EuroQoI-5D-5L)
* Supra-gingival polishing and reinforcement of oral hygiene instructions

Visit 8 - 6 months follow up visit- (6 months ±7 days from visit 2)

* Query to update medical/dental history and record adverse events and/or concomitant medications
* Recording of PPD, REC, BOP, PI and mobility on the tooth involved in the surgical intervention and 2 adjacent teeth by a blind and calibrated examiner
* Supra-gingival polishing and reinforcement of oral hygiene instructions
* PROMsS assessment (OIDP, Global ratings of Periodontal Health and Quality of Life, and eEvaluation of global changes in quality of life and EuroQoI-5D-5L)

Visit 9 - 12 months follow up visit- (12 months ±7 days from visit 2)

* Query to update medical/dental history and record adverse events and/or concomitant medications
* Periodontal assessment by a blind and calibrated examiner, consisting of full mouth PPD, REC, BOP, mobility and furcation involvement will be recorded. PPD, REC, plaque and BOP will be recorded at 6 sites per tooth.
* PROMS assessment (OIDP, Global ratings of Periodontal Health and Quality of Life, and eEvaluation of global changes in quality of life and EuroQoI-5D-5L)
* Supra-gingival polishing and reinforcement of oral hygiene instructions
* Standardised peri-apical x-ray in the area selected for the study

Study randomisation and treatment allocation Following completion of the preparation treatment all individuals enrolled into the study will be randomly assigned to one of the treatment groups.

* Simplified Papilla Preservation Flap (SPPF) and guided tissue regeneration (GTR) with a porcine collagen membrane and a deproteinized bovine bone substitute.
* Simplified Papilla Preservation Flap (SPPF) and PRGF ENDORET.

A balanced random permuted block approach (4-unit block size) will be used to prepare the randomisation tables. Minimisation will be carried out to facilitate balancing of smokers in each group.

Allocation to treatment will take place via the study coordinator (or one of their delegate). Treatment allocation details will be concealed in an opaque envelope at the study site.

At the time of enrollment, each participant will be sequentially issued a subject ID. The subject ID consists of two initials and a number. The ID number will consist of three digits and will be assigned in ascending numerical order beginning with 001.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy males and females ≥25 years old
* Willingness to read and sign a copy of the Informed Consent Form after reading the Patient Information Sheet, and after the nature of the study has been fully explained
* Clinical evidence of periodontitis, with one interdental area of PPD ≥6mm, BOP, and attachment loss ≥6mm, with associated intrabony defect ≥3mm in any area of their mouth (excluding third molars and distal of second molars)
* Full mouth bleeding and plaque scores (FMBS and FMPS) <25%recorded within the previous 6 weeks
* Non-surgical treatment completed within 6 months prior to assessment for eligibility

Exclusion Criteria:

* Medical history that includes diabetes type 1 or hepatic or renal disease, or other serious medical conditions or transmittable diseases (e.g. cardiovascular disease or AIDS).
* Antibiotic or anti-inflammatory therapy during the month preceding the baseline exam.
* In chronic treatment (>2 weeks) with anticoagulants, corticosteroids or other medications that can severely impact on bone formation
* History of alcohol or drug abuse.
* Smoking ≥10 cigarettes a day
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing, which can affect interpretation of study results).
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgement of the investigator, would make the subject inappropriate for entry into this trial.
* Periodontal surgery in the same area selected for the study within the past 12 months.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changed in Probing Pocket Depth (PPD) | 12 months after treatment
  Changes in PPD from baseline to 12 months after treatment

SECONDARY OUTCOMES:
Patients' reported outcomes (PROMs) in Oral Impact on Daily Performances (OIDP) questionnaire (OIDP). | At baseline, 3 months after surgery (visits 2), 6 months after surgery, 12 months after surgery.
  The OIDP is a well validated and frequently used PROM in studies of oral health. It is a composite measure of the impacts of oral health on the quality of life of people. The OIDP focuses on the impact that the conditions of the teeth and mouth have on the physical (functional), psychological and social wellbeing of the person. More specifically, it assesses the impact of oral conditions on basic daily life activities and behaviours (eating, speaking, cleaning teeth, going out, relaxing, smiling, major work or role, emotional stability, social contact). For each performance, both the frequency and severity of oral impacts are assessed. The overall OIDP score ranges from 0 to 100, with higher scores indicating worse quality of life.
PROMs based on Global ratings of Periodontal Health and Quality of Life | At baseline, 4 weeks after surgery (visit 2), 3 months after surgery, 6 months after surgery, 12 months after surgery.
  PROMs based on Global ratings of Periodontal Health and Quality of Life
PROMs based on the evaluation of global changes in quality of life | At baseline, 2 days after surgery (visit 2), 7 days after surgery, 14 days after surgery, 4 weeks after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery.
  Global ratings on health and quality of life will be provided through two methods:
  a) the Visual Analogue Scale (VAS) included in the EQ5D questionnaire. b) through the following question: 'How would you rate the quality of your life'?
  The responses will be scored on a six-point scale as:
  1. Excellent
  2. Very good
  3. Good
  4. Fair
  5. Poor
  6. Very poor
  PROMs based on the evaluation of global changes in quality of life;
PROMs based on the evaluation of patient perception about therapy | At baseline, 2 days after surgery (visit 2), 7 days after surgery, 14 days after surgery, 4 weeks after surgery.
  The extent of discomfort and/or pain experienced will be evaluated using a 100-mm horizontal visual analog scale (VAS). The anchors for each end of the scales will be designated as none and extreme. Patients will be also instructed to quantify the analgesic medication taken. In addition, the extent of discomfort, root hypersensitivity, oedema, hematoma, high fever, and interference in daily activities during the first post-therapy week will be evaluated in the same way.
Post-operative swelling and oedema | At baseline, within 6 weeks from baseline (at visit 2 - surgical intervention), 2, 7 and 14 days after surgical intervention (visit 2)
  A series of subtracted images from the baseline will accurately identify the area and magnitude of the swelling, changes in facial shape, volume and temperature to monitor/quantify the healing. For every patient, a person specific template of postoperative facial swelling/ oedema pattern will be created for sequential swelling/thermal changes or oedema volume measurements that will be applied on a unique alignment of the patient's specific consecutive imaging surfaces (self- defined positioning based on patient's facial features).
Changes in blood flow | At baseline and 2, 7 and 14 days after surgical intervention (visit 2)
  The vascularization pattern of the peri-implant soft tissues will be evaluated with Laser Speckle Contrast Imaging (LSCI), according to the methodology described by previous studies. LSCI is a radiation-free, non-invasive procedure to assess blood flow. Systolic and diastolic blood pressure as well as pulse rate will be measured with an automatic blood pressure monitor before and after the LSCI measurements. These measures will be combined to give a measure of blood flow to assess patients' vascularization pattern of the peri-implant soft tissues. Each patient will seat comfortably in supine position in a dental chair, and a vacuum pillow will be used for fixing their head. The patient will be left undisturbed for 15 minutes before any measurements will be taken. All measurements will be carried out at a constant room temperature.
Radiographic bone changes | From baseline to 12 months post-surgery
  Standardised intraoral radiographs will be taken on the tooth involved in the surgical intervention at baseline and at 12 months post treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Barts and The London Dental Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No